CLINICAL TRIAL: NCT03620019
Title: Phase 2 Study of Denosumab in Combination With a PD-1 Inhibitor in Subjects With Stage III/IV Melanoma
Brief Title: Denosumab + PD-1 in Subjects With Stage III/ IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1620
Record Dates: First submitted 2018-07-11; First posted 2018-08-08 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Melanoma Stage Iii; Melanoma Stage Iv; Melanoma; Melanoma (Skin); Cutaneous Melanoma
Keywords: Denosumab; Pembrolizumab; Melanoma; Unresectable; Cutaneous; Nivolumab
MeSH Terms: conditions — Melanoma | interventions — Denosumab; pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm: Denosumab+ PD-1 Inhibitor (Experimental): Subjects in this trial will be given denosumab every 4 weeks, starting on day 1 of study treatment. An additional loading dose of denosumab will be administered on day 8. Subjects who started Pembrolizumab (initiated 21 days after the first dose of denosumab is given) will continue to have it administered intravenously (IV) every 3 weeks. New subjects will receive Nivolumab administered intravenously (IV) every 4 weeks (initiated 21 days after the first dose of denosumab is given). Combination therapy will continue as long as subjects benefit from therapy for up to 1 year.
  Interventions: Drug: Denosumab; Drug: Pembrolizumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Denosumab — A dose of 120 mg will be administered as a subcutaneous (s.c.) injection every 4 weeks in the upper arm, upper thigh, or abdomen. Another loading dose of 120 mg s.c. denosumab will be administered on day 8. On days when denosumab is administered on the same day as pembrolizumab, the s.c. injection should be given after the infusion of pembrolizumab is completed.
  Other Names: XGEVA
Drug: Pembrolizumab — Pembrolizumab will be administered as standard of care following the institutional guidelines.The recommended dose of pembrolizumab is 200 mg administered as an IV infusion over approximately 30 minutes (range: 25 - 40 minutes) every 3 weeks until disease progression or unacceptable toxicity.
  Other Names: Keytruda
Drug: Nivolumab — Nivolumab will be given every four weeks at a dose of 480 mg to be administered as an IV infusion per institutional guidelines.
  Other Names: Opdivo

SUMMARY:
This is a multicenter open-label, single-arm, phase II study designed to investigate the pharmacodynamic and antitumor effects of denosumab alone and in combination with an anti-Programmed death-1 or Programmed death ligand 1 (PD1) agent (pembrolizumab or nivolumab) in patients with unresectable Programmed death-1 or Programmed death ligand 1 (PD-1/PD-L1) inhibitor-naïve regional and distant metastatic melanoma (The American Joint Committee on Cancer (AJCC) stage III/IV). The pharmacodynamic and antitumor effects will be investigated by performing translational research on peripheral blood and tumor tissue collected before and during denosumab alone and in combination with anti-PD-1 treatment.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Co-primary Objectives

* Assess the mechanistic (immune-mediated and/or direct antitumor effect) and pharmacodynamics effect (tissue saturation studies) of denosumab alone (i.e., after three loading doses of denosumab are given on days 1,8 and 22) in patients with unresectable (or resectable) stage III or distant metastatic PD-1/PD-L1 inhibitor-naïve cutaneous melanoma (stage III/IV) by performing translational research on peripheral blood and tumor biopsy samples collected at baseline and after third loading dose of Denosumab.
* Assess the immune-mediated and direct antitumor effect of denosumab in combination with anti- PD-1 agent in patients with unresectable (or resectable) stage III or distant metastatic PD-1/PD-L1 inhibitor-naïve cutaneous melanoma (The American Joint Committee on Cancer (AJCC) stage III/IV) by performing translational research on peripheral blood and tumor biopsy samples collected at weeks 16, 28 and 40 of the study and comparing the results with those from baseline and after third loading dose of Denosumab.

Secondary Objectives

* Assess the safety of the denosumab-anti-PD-1 agent combination in unresectable (resectable) stage III or distant metastatic PD-1/PD-L1 inhibitor-naïve melanoma (The American Joint Committee on Cancer (AJCC) stage III/IV) by National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
* Determine antitumor response by Response evaluation criteria in solid tumors (RECIST) v1.1 criteria of the denosumab-anti- PD-1 agent combination at 16 weeks in patients with unresectable (resectable) stage III or distant metastatic PD-1/PD-L1 inhibitor-naïve melanoma (The American Joint Committee on Cancer (AJCC) stage III/IV).
* Determine the 1-year Overall Survival rate of the Denosumab-anti-PD-1 agent combination in patients with unresectable (or resectable) stage III or distant metastatic PD-1/PD-L1 inhibitor-naïve melanoma (The American Joint Committee on Cancer (AJCC) stage III/IV).
* Determine the 6-month PFS rate of the denosumab-anti-PD-1 agent combination in patients with unresectable (or resectable) stage III or distant metastatic PD-1/PD-L1 inhibitor-naive melanoma (The American Joint Committee on Cancer (AJCC) stage III/IV).

Endpoints Co-primary Endpoints

* The immune-mediated mechanism of action of denosumab alone will be evaluated in blood and tumor samples collected at baseline and after the third loading dose of denosumab. Multiparameter flow cytometry and ELISA assays will be performed on peripheral blood/serum samples as outlinedin the protocol. Tumor biopsy samples will be evaluated by IHC and IF studies as outlined in the protocol.
* The immune-mediated mechanism of action of denosumab combined with anti-PD-1 agent will be evaluated in blood and tumor samples collected at weeks 16, 28, and 40 of the study. Multi-parameter flow cytometry and ELISA assays will be performed on peripheral blood/serum samples collected at weeks 16, 28, and 40 as outlined in the protocol. Tumor biopsy samples obtained at week 16 will be evaluated by immune histochemical (IHC) and immune florescent (IF) studies as outlined in the protocol.

Secondary Endpoints

* Adverse Events (AE) experienced by patients receiving denosumab-anti- PD-1 agent will be assessed per National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
* The overall response (complete response + partial response ) at 16 weeks will assessed based on Response evaluation criteria in solid tumors (RECIST) v1.1 criteria.

The overall Survival (OS) rate at 1 year is defined as the time from day 1 of study treatment until death as a result of any cause within one year of initiating study treatment.

-Progression Free Survival (PFS) rate at 6 months is defined as the time from day 1 of treatment until disease progression or death status measured 6 months after initiating study treatment. Progression events will be defined per Response evaluation criteria in solid tumors (RECIST) v1.1 criteria.

Procedures

Subjects in this trial will be given denosumab, 120 mg s.c. q4 weeks, starting on day 1 of study treatment. Additional loading doses of Denosumab will be administered on day 8 and day 22 ( after Amendment 1). Nivolumab, 480 mg will be administered intravenously (IV) every 4 weeks and initiated 21 days after the first dose of Denosumab is given. In subjects enrolled prior to Amendment 1 Pembrolizumab, 200 mg will be administered intravenously (IV) every 3 weeks and initiated 21 days after the first dose of denosumab is given. Combination therapy with both agents will continue as long as subjects benefit from therapy for up to 1 year. Study therapy will be discontinued for intolerable toxicity, disease progression or for other reasons at the discretion of the investigator. If subjects are not withdrawn prematurely then their last dose of study medications will be administered approximately 49 weeks after denosumab was initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent and HIPAA authorization for release of personal health information.
2. Age ≥ 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
4. Histologically confirmed melanoma of cutaneous or mucosal primary; (e.g. sinus, vagina, anus, gastrointestinal tract); metastatic melanomas from unknown primary are allowed because melanoma of unknown primary is biologically similar to cutaneous melanomas.
5. AJCC stage III/IV unresectable (or resectable) disease. Both should be measurable by RECIST v1.1 criteria. Patients with resectable bulky stage IIIB, state IIIC or stage IIID melanoma (≥2-cm in shortest diameter for lymph nodes infiltrated by tumor and ≥2-cm in longest diameter for non-lymph nodes infiltrated by tumor) can also be entered into the study at the discretion of the Principal Investigator.
6. Must have available and consent to collect archived tumor blocks from previous surgeries confirming or treating metastatic disease (e.g. radical lymph node dissection); if not available they can be enrolled into the trial, if they consent to have a tumor biopsy before treatment initiation.
7. Must agree to undergo one on-treatment biopsy on week 4of the study; the biopsy at week 16 is optional.
8. Must agree to have 100 mL blood drawn for study purposes on week 1 , day 20+or-2 (week 4), week 16, week 28, week 40 and end of treatment.
9. Demonstrate adequate organ function, as listed below; all screening labs are to be obtained within 21 days prior to registration.

   * Hemoglobin ≥ 10 g/dL without transfusion or erythropoietin dependency (within 7 days of assessment)
   * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   * Absolute Lymphocyte Count (ALC) ≥ 1,000/mm3
   * Platelets≥ 100,000/mm3
   * Serum Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 × upper limits of normal (ULN) OR
   * ≥ 60 mL/min using the Cockcroft-Gault formula for subjects with creatinine levels > 1.5 × ULN
   * Serum Total Bilirubin ≤ 1.5 × ULN or ≤ 2 × ULN for subjects with Gilbert's Syndrome
   * Aspartate aminotransferase (AST) ≤ 2.5 × ULN OR < 5 × ULN for subjects with liver metastases
   * Alanine aminotransferase (ALT) ≤ 2.5 × ULN OR < 5 × ULN for subjects with liver metastases
   * Albumin ≥ 2.5 mg/dL
   * Serum calcium ≥ 2.0 mmol/L (8.0 mg/dL)
10. Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to study treatment. Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
11. Females of childbearing potential must be willing to use an adequate methods of contraception, as outlined in the protocol. Oral contraception is required 14 days prior to initiation of study medications until 120 days after treatment discontinuation. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception as outlined in the protocol- Contraception, starting with the first dose of study therapy through 150 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
13. As determined by the enrolling physician or protocol designee, willingness and ability of the subject to understand and comply with study procedures.
14. Previous radiation therapy is allowed, provided it is completed ≥14 days prior to starting denosumab and patient has recovered adequately from any related toxicities (grade≤1, or grade ≤2 that is stable for ≥3 months).
15. If patient has received adjuvant treatments, in particular ipilimumab and high dose interferon, any toxicities must have resolved to grade 1 or less. Grade 2 toxicities attributed to ipilimumab from autoimmune endocrinopathies that require permanent hormone replacement therapy are allowed as long as they are adequately treated. This implies that patients should be off systemic steroids for treatment of any of these or other autoimmune toxicities (e.g. colitis, rash).

Subjects who have previously received PD-1 inhibitors in stage III (adjuvant) or stage IV are allowed as long as:

1. the interval between the last dose of the adjuvant PD-1 inhibitor and the date of relapse (clinical or radiographic) is at least 1 year,
2. if subjects who received treatment for stage IV had antitumor response (partial response or complete response) by RECIST criteria version 1.1 but they stopped due to subject/investigator preference for at least a year between the last dose of the PD-1 inhibitor and the date of relapse (clinical or radiographic). Allowing for these subjects who have previously received PD-1 inhibitors in the adjuvant setting (i.e. no knowledge about clinical benefit) or following definite antitumor response in the metastatic setting is based on a recent case series of subjects who responded to PD-1 inhibitor rechallenge, if they had previously responded to PD-1 inhibitors. This implies that waning antitumor immunity in the absence (i.e. >1 year) of costimulation with PD-1 inhibitors may be the reason for cancer recurrence and NOT primary resistance of PD-1 inhibitors.
3. any side effects that may have occurred during the previous exposure to PD-1 inhibitors are not serious (i.e. grade 1 or 2 by CTCAE version 5.0 criteria).

Exclusion Criteria:

1. History of prior malignancy, with the exception of the following:

   * Non-melanoma skin cancers, non-invasive bladder cancer, and carcinoma in situ of the cervix,
   * Prior history of prostate, provided that patient is not under active systemic treatment other than hormonal therapy and with documented undetectable prostate specific antigen (PSA < 0.2 ng/mL),
   * Chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) provided patient has isolated lymphocytosis (Rai stage O), and does not require systemic treatment [for "B" symptoms, Richter's transformation, lymphocyte doubling time (< 6 months), lymphadenopathy or hepatosplenomegaly],
   * Lymphoma or any type or hairy-cell leukemia, provided patient is not on an active systemic treatment and is in complete remission, as evidenced by Positron Emission Tomography (PET)/CT scans and bone marrow biopsies for at least 3 months,
   * History of other malignancy, provided patient has completed therapy, or does not require therapy, and is free of disease for ≥ 2 years. If patient has had other malignancy within the last 2 years from which he/she may have been completely cured by surgery alone, or does not require any treatment other than observation at the specialist's discretion, he/she may considered to be enrolled on condition that the risk of development of recurrent or distant metastatic disease based on the American Joint Committee in Cancer (AJCC) staging system is less than 30% in 3 years from the original diagnosis of other malignancy.
2. Has known active central nervous system (CNS) metastases that are symptomatic and require antiepileptic drugs or corticosteroids (any dose). Subjects with previously treated brain metastases may participate provided they are asymptomatic (i.e., no neurologic symptoms) for at least 2 weeks prior to the first dose of trial treatment and are not using steroids for at least 7 days prior to trial treatment. Patients with previously treated brain metastases should have evidence of stable brain metastases (without evidence of progression by imaging) for at least 2 weeks prior to the first dose of trial treatment. Patients with previously treated but grown brain metastases (or new brain metastases if there is no prior history of brain metastases) are still allowed in the study as long as the net growth of pre-existing brain lesions (or new brain lesions if there is no prior history of brain metastases) does not exceed 1-cm in largest diameter as measured by brain MRI with IV contrast (for example, a patient with pre-existing brain lesion(s) that has grown by 6-mm in the largest diameter and also has a new lesion that measures 4-mm in largest diameter can still be enrolled in the study; alternatively, a patient that has a new brain lesion that measures 1-cm in the largest diameter and no growth of pre-existing brain lesions can still be enrolled in the study). This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability. Subjects with leptomeningeal disease, detected either by brain MRI or by cytology (e.g. lumbar puncture) are also excluded.
3. Treatment with any investigational drug, immunotherapy or chemotherapy within 28 days prior to study treatment (i.e., initiation of denosumab). Treatment with any targeted therapy (e.g. Mitogen-Activated Protein Kinases (MAPK) inhibitors) is allowed as long as at least 15 days have elapsed since last dose of drug.
4. Patients discontinuing prior therapy with tyrosine kinase inhibitors for melanoma should be off these medications for at least 15 days before starting study treatment.
5. Prior PD-1/PD-L1 therapies in the adjuvant setting; targeted therapies or prior ipilimumab in the adjuvant setting are allowed.
6. Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk, if he/she were to participate in the study. This includes, but is not limited, to serious medical conditions or psychiatric illness likely to interfere with participation in this clinical study.
7. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy equivalent to daily doses of prednisone of 10 mg or greater (or an equivalent dose of other corticosteroids) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
8. Has a known history of active tuberculosis (Mycobacterium Bacillus Tuberculosis).
9. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
10. Hypersensitivity to nivolumab, pembrolizumab or denosumab or any of their excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of non-infectious pneumonitis that required systemic corticosteroids or evidence of interstitial lung disease or current active, non-infectious pneumonitis Episodic, brief (< 7 day) exposure to systemic corticosteroids (e.g. steroid taper for poison ivy or chronic obstructive pulmonary disease (COPD) exacerbation) is allowed.
13. Has a history of an acute coronary event (e.g. myocardial infarction) within 3 months since study entry, uncontrolled and symptomatic coronary artery disease, or congestive heart failure New York Heart Association class III/IV.
14. Has an active infection requiring systemic therapy within 7 days prior to treatment initiation.
15. Has a known history of Human Immunodeficiency Virus (HIV 1/2 antibodies).
16. Known serologic status reflecting active hepatitis B or C infection. Patients that are hepatitis B core antibody positive, but antigen negative, will need a negative polymerase chain reaction (PCR) prior to enrollment. [Note: Hepatitis B antigen or PCR positive patients will be excluded].
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.
18. Known active metabolic bone disease such as Paget's disease, Cushing's disease, hyperprolactinemia, over the last year 12 months, known history of osteoporosis that is symptomatic (e.g. history of fractures, bone pain), or hypercalcemia/hypocalcemia of any type (serum-free calcium being more than 1.1 x upper limit of normal (ULN) and less than 0.9 x, lower limits normal. LLN) over the last 2 weeks since study initiation that requires treatment beyond calcium and vitamin D supplementation.
19. Prior treatment with denosumab. Use of bisphosphonates for the treatment of metastatic bone disease, but not for hypercalcemia of malignancy, is allowed.
20. History of current evidence of osteonecrosis or osteomyelitis of the jaw. Note: The subject should be referred to dentist before study treatment initiation for poor dentition or other dental issues that, in the opinion of the treating physician, may increase the risk of osteonecrosis of the jaw.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Moschos, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Manchester, New Hampshire
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-five subjects were enrolled in the study between 09/10/2018-05/31/2022 in 2 centers in the United States.
Period: Overall Study
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects started to the study treatment.
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.12 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: The Antitumor Effect of Denosumab Alone as Represented by the Change in Recent Thymic Emigrant Cells in Peripheral Blood
Description: The antitumor effect of denosumab alone (i.e., after two loading doses of denosumab are given on day 1 and day 8) in patients with unresectable stage III or distant metastatic Programmed death-1 or Programmed death ligand 1 (PD-1/PD-L1) inhibitor-naïve cutaneous melanoma (stage III/IV) will be assessed by performing translational research on peripheral blood samples collected at baseline and on day 21 of the study. The hypothesis is that denosumab treatment will prevent the destruction of autoreactive T cells within the thymus -and therefore will increase the influx of those T cells into the blood, termed recent thymic emigrants (RTE). RTE will be measured by multiparameter flow cytometric analysis of cluster of differentiation CD4+ and CD8+ RTE isolated from peripheral blood. Results will be expressed as the change in the number of cells/microliter of peripheral blood between the baseline and the day 21 time points.
Time Frame: 3 weeks after start of denosumab
Population: Subjects received denosumab alone and provided blood sample at baseline and week 3.
Measure: Mean (Full Range); unit: number of cell per microliter
Groups:
- CD4+ Baseline: CD4+ values were determined from peripheral blood samples collected at baseline.
- CD8+ Baseline: CD8+ values were determined from peripheral blood samples collected at baseline
- CD4+ at 3 Weeks: CD4+ values were determined from peripheral blood samples collected at 3 weeks of the study.
- CD8+ at 3 Weeks: CD8+ values were determined from peripheral blood samples collected at 3 weeks of the study.
Arm/Group | CD4+ Baseline | CD8+ Baseline | CD4+ at 3 Weeks | CD8+ at 3 Weeks
Number analyzed (Participants) | 23 | 23 | 23 | 23
number of cell per microliter | 2.69 [0.34 to 15.9] | 2.42 [0.34 to 15.9] | 2.55 [0.32 to 12] | 1.92 [0.32 to 12]

2. Primary Outcome: The Antitumor Effect of Denosumab Alone as Represented by the Change in Density of Tumor-infiltrating Cluster of Differentiation (CD8+) Cells (TILs) in Tumor Tissue.
Description: The antitumor effect of denosumab alone (i.e., after two loading doses of denosumab are given on day 1 and day 8) in patients with unresectable stage III or distant metastatic Programmed death-1 or Programmed death ligand 1 (PD-1/PD-L1) inhibitor-naïve cutaneous melanoma (stage III/IV) will be assessed by performing translational research on tumor biopsy samples collected at baseline and on day 21 of the study. The hypothesis is that denosumab alone will increase influx of tumor-infiltrating CD8+ cells (TIL). The density of TILs (number of cells by tumor surface area in mm2) in tumor tissues will be evaluated by Immunohistochemistry (IHC) and Immunofluorescence (IF) studies.
Time Frame: 3 weeks after start of denosumab
Population: Subjects who started Denosumab alone study treatment, tumor-infiltrating Cluster of Differentiation (CD8+) Cells (TILs) in Tumor Tissue tests were performed at baseline and on day 21, were included. Although a biopsy was taken from all the subjects, tissue samples of 4 subjects were not included due to no presence of viable tumors or a necrotic tumor was present.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 20
Participants
  The number of subjects with TIL values decreased | 9
  The number of subjects with TIL values stable | 7
  The number of subjects with TIL values increased | 4

3. Primary Outcome: The Antitumor Effect of Denosumab Combined With Anti-PD-1 Inhibitor as Represented by the Change in Recent Thymic Emigrant Cells in Peripheral Blood - CD8+
Description: The antitumor effect of denosumab combined with anti-PD-1 inhibitor (Pembrolizumab or Nivolumab) in patients with unresectable stage III or distant metastatic Programmed death-1 or Programmed death ligand 1 (PD-1/PD-L1) inhibitor-naïve cutaneous melanoma (stage III/IV) will be assessed by performing translational research on peripheral blood samples collected at weeks 16, 28 and 40 of the study. The hypothesis is that denosumab treatment will prevent the destruction of autoreactive T cells within the thymus -and therefore will increase the influx of those T cells into the blood, termed recent thymic emigrants (RTE). RTE will be measured by multiparameter flow cytometric analysis of cluster of differentiation (CD)8+ and CD 4+ RTE isolated from peripheral blood. Results will be expressed as the change in the number of cells/microliter of peripheral blood between the week 16, 28, and 40 time points.
Time Frame: 16, 28 and 40 weeks after start of denosumab
Population: Subjects received denosumab combined with anti-PD-1 inhibitor (Pembrolizumab or Nivolumab) and provided blood samples at weeks 16, 28, and 40.
Measure: Mean (Full Range); unit: valuenumber of cell per microliter
Groups:
- CD4+ Week 16: CD4+ values were determined from peripheral blood samples collected at week16.
- CD8+ week16: CD8+ values were determined from peripheral blood samples collected at week 16.
- CD4+ at Week 28: CD4+ values were determined from peripheral blood samples collected at week 28.
- CD8+ at Week 28: CD8+ values were determined from peripheral blood samples collected at week 28.
- CD4+ at Week 40: CD4+ values were determined from peripheral blood samples collected at week 40.
- CD8+ at Week 40: CD8+ values were determined from peripheral blood samples collected at week 40
Arm/Group | CD4+ Week 16 | CD8+ week16 | CD4+ at Week 28 | CD8+ at Week 28 | CD4+ at Week 40 | CD8+ at Week 40
Number analyzed (Participants) | 23 | 23 | 15 | 15 | 13 | 13
valuenumber of cell per microliter | 2.06 [0.06 to 7.58] | 1.64 [0.06 to 7.58] | 2.84 [0.16 to 20.3] | 2.76 [0.16 to 20.03] | 2.27 [0.4 to 11] | 1.76 [0.4 to 11]

4. Primary Outcome: The Antitumor Effect of Denosumab Combined With Anti-PD-1 Inhibitor as Represented by the Change in Density of Tumor-infiltrating Cluster of Differentiation (CD8+) Cells (TILs) in Tumor Tissue.
Description: The antitumor effect of denosumab combined with anti-PD-1 inhibitor (Pembrolizumab or Nivolumab) in patients with unresectable stage III or distant metastatic Programmed death-1 or Programmed death ligand 1 (PD-1/PD-L1) inhibitor-naïve cutaneous melanoma (stage III/IV) will be assessed by performing translational research on tumor biopsy samples collected at baseline, on day 21, and week 16 of the study. The density of TILs (number of cells by tumor surface area in mm2) in tumor tissues will be evaluated by Immunohistochemistry (IHC) and Immunofluorescence (IF) studies.
Time Frame: Baseline, 16 weeks after start of denosumab combined with anti-PD-1 inhibitor
Population: Subjects who started study treatment, Denosumab Combined With Anti-PD-1 Inhibitor, Tumor-infiltrating Cluster of Differentiation (CD8+) Cells (TILs) in Tumor Tissue tests were performed, at baseline and 16 weeks after the treatment were included. Biopsy on week 16 was not mandatory per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 3
Participants
  The number of subjects with TIL value decreased between week 3 to week 17 | 0
  The number of subjects with TIL value increased between week 3 to week 17 | 3

5. Secondary Outcome: Number of Participants With Treatment-related Serious Adverse Events of the Denosumab Alone Plus Its Combination With Nivolumab
Description: The safety of the denosumab- anti-PD-1 inhibitor (Pembrolizumab or Nivolumab) combination will be assessed by continuous toxicity monitoring focusing on the incidence of serious adverse events (SAEs) with toxicity boundary rules. The NCI Common Terminology Criteria for Adverse Events V5 is a descriptive terminology which will be used for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 30 days after treatment is discontinued
Population: Subjects received the study treatment and adverse events were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 25
Participants
  Rash maculo-papular | 1
  Pneumonitis | 1
  Colitis | 1

6. Secondary Outcome: Overall Response Rate
Description: Antitumor response to the denosumab- anti-PD-1 inhibitor (Pembrolizumab or Nivolumab) combination at 16 weeks in patients with unresectable stage III or distant metastatic PD-1/PD-L1 inhibitor-naïve cutaneous melanoma (AJCC stage III/IV) will be assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) which defines Complete Response (CR) as Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Overall Response Rate (ORR) = CR + PR/total number of subjects.
Time Frame: 16 weeks after start of treatment
Population: Subjects received the study treatment and tumor response were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 17
Participants
  Complete Response | 2
  Partial Response | 5
  Stable | 5
  Progression | 5

7. Secondary Outcome: Overall Survival Rate
Description: The Overall Survival rate at 1-year is defined as the proportion of subjects still alive from day 1 of study treatment until one year after initiating study treatment
Time Frame: 1 year from start of study treatment
Population: Subjects received the study treatment and were followed-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 23
Participants
  Alive | 18
  Died | 5

8. Secondary Outcome: Progression Free Survival Rate
Description: Progression Free survival rate at 6 months is defined as the proportion of subjects without a progression or death event measured from day 1 of treatment until 6 months after initiating study treatment. Progression events will be defined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 months from start of study treatment
Population: Subjects received the study treatment and tumor responses were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
Number analyzed (Participants) | 23
Participants
  Progression | 11
  No progression | 12

ADVERSE EVENTS:
Time Frame: Up to 56 weeks
Description: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment. Any hospital admission was graded as a serious adverse event per protocol.
Arm/Group | Single Arm: Denosumab+ PD-1 Inhibitor
All-Cause Mortality (participants affected / at risk) | 5/25
Serious Adverse Events (participants affected / at risk) | 13/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: Denosumab+ PD-1 Inhibitor (N=25)
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Lymphocyte count decreased (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: Denosumab+ PD-1 Inhibitor (N=25)
Anemia (Blood and lymphatic system disorders) | 6
Eosinophilia (Blood and lymphatic system disorders) | 4
Lymph node pain (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 4
Testosterone deficiency (Endocrine disorders) | 5
Blurred vision (Eye disorders) | 3
Cataract (Eye disorders) | 1
Dry eye (Eye disorders) | 6
Eye disorders - Other, specify (Eye disorders) | 2
Floaters (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 14
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Gingival pain (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Stomach pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Eye disorders) | 2
Chills (General disorders) | 2
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 20
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 5
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 11
Allergic reaction (Immune system disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 3
fall (Injury, poisoning and procedural complications) | 1
fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 6
Blood bicarbonate decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 4
Blood prolactin abnormal (Investigations) | 1
Creatinine increased (Investigations) | 2
Hemoglobin increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 4
Lipase increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Serum amylase increased (Investigations) | 4
Thyroid stimulating hormone increased (Investigations) | 4
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Muscle cramp (Musculoskeletal and connective tissue disorders) | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 11
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 8
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 2
Glucosuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 11
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 4
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03620019/Prot_SAP_000.pdf